CLINICAL TRIAL: NCT05902884
Title: New Biomarkers in Facioscapulohumeral Muscular Dystrophy, Multispectral Optoacoustic Tomography.
Acronym: MSOT-FSHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5374
Record Dates: First submitted 2023-04-27; First posted 2023-06-15 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-04

CONDITIONS: FSHD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Patients with FSHD
  Interventions: Device: MSOT Acuity Echo
- Controls (Other): Healthy volunteers
  Interventions: Device: MSOT Acuity Echo

INTERVENTIONS:
Device: MSOT Acuity Echo — Imaging of muscles applying Multi-spectral optoacoustic tomography (MSOT)

SUMMARY:
Facioscapulohumeral Muscular Dystrophy (FSHD) is one of the most frequent muscular dystrophies in the adulthood. Multi-spectral optoacoustic tomography (MSOT) is an innovative imaging technique able to non-invasively characterize the molecular composition of the muscle tissue. With this pilot study we will explore the performance of MSOT imaging in FSHD patients and correlate the findings with clinical and MRI data, with the final aim to identify new disease biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* molecular diagnosis of FSHD
* recent pelvic and lower-limb muscle MRI

Exclusion Criteria:

* presence of conditions that can alter the signal of the muscles under investigation: eg. tattoos, scars or skin abrasions at the site of probe evaluation, recent trauma, decompensated diabetes, symptomatic radiculopathies, acute or chronic inflammatory diseases
* current or presumed pregnancy
* inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Optoacoustic Absorption Spectrum (peaks at different wavelengths in arbitrary units) in FSHD muscles | 6 months
  Definition of the Optoacoustic Absorption Spectrum (glycogen, lipid, collagen, hemo/myoglobin peaks at different wavelengths in arbitrary units) of muscles of FSHD patients and evaluation of the differences compared to healthy volunteers.

SECONDARY OUTCOMES:
Medical Research Council (MRC) Muscle Strength Grades | 6 months
  Correlation of spectra detected by MSOT with clinical scores
Disease severity (Clinical Severity Scale CSS) | 6 months
  Correlation of spectra detected by MSOT with Clinical Severity Scale(CSS), a global index of disease severity specific for FSHD (from 0 to 5 points).
Phenotyping (FSHD Comprehensive Clinical Evaluation Form CCEF) | 6 months
  Correlation of spectra detected by MSOT with the phenotype classification derived applying the FSHD Comprehensive Clinical Evaluation Form CCEF (4 categories)
Dynamometer test of muscle strength | 6 months
  Correlation of spectra detected by MSOT with muscle strength (in N) assessed using a hand held dynamometer
Magnetic resonance imaging | 6 months
  Correlation of spectra detected by MSOT with magnetic resonance imaging parameters (presence of fatty replacement in T1-weighted sequences, presence of increased signal in short-tau inversion recovery sequences)
Intraclass correlation coefficient | 6 months
  Evaluation of intra and inter-observer agreement in the estimate of Optoacoustic Absorption Spectra using Intraclass correlation coefficient (ICC) of the repeated measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy